CLINICAL TRIAL: NCT04900636
Title: A Telemedicine Platform for Patients With Type 1 Diabetes Mellitus Treated With an Hybrid Closed Loop System
Brief Title: Telemedicine for Patients With an Hybrid Closed Loop System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 317/19
Record Dates: First submitted 2021-05-18; First posted 2021-05-25 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Arm (Experimental): Use of a telemedicine platform combined with face-to-face visits according to protocol
  Interventions: Device: Telemedicine Arm
- Control Arm (No Intervention): conventional follow-up according to routine clinical practice.

INTERVENTIONS:
Device: Telemedicine Arm — Patients with DM1 ≥ 18 years of age, users of closed loop hybrid systems, assigned to a follow-up program using a telemedicine platform combined with face-to-face visits according to protocol.
  Arms: Telemedicine Arm

SUMMARY:
The primary objective is to assess the impact on quality of life after a follow-up program using a telemedicine platform designed for patients with DM1 treated with an hybrid closed loop insulin infusion system. Open-label, randomized 1:1 controlled clinical trial during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for DM1 according to ADA
* They must have access to the technology that allows monitoring (mobile phone and / or computer as well as having an internet connection)
* Acceptance of participation in the study and signing of the informed consent

Exclusion Criteria:

* Gestation
* Institutionalization, serious or terminal illness or renal replacement therapy.
* Inability to undertake the training and / or acquire the degree of knowledge to use the telemedicine platform.
* Refusal to participate in the study or to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Impact on quality of life | 12 months
  Health-related quality of life in patients with type 1 diabetes (the ViDa1 questionnaire). The four-dimensional structure for ViDa1 are:
  * Interference of diabetes in everyday life (the minimum value: 12 and maximum value: 60) higher scores mean a worse outcome
  * Self-care (the minimum value: 11 and maximum value: 55) higher scores mean a better outcome
  * Well-being (the minimum value: 6 and maximum value: 30) higher scores mean a better outcome, and
  * Worry about the disease (the minimum value: 5 and maximum value: 25) higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Metabolic control | 12 months
  A1c levels

CONTACTS AND LOCATIONS:
Overall Officials: Lía Nattero Chávez, MD PhD, Principal Investigator — Hospital Ramón y CajaDiabetes, Obesity and Human Reproduction Research Group, Department of Endocrinology and Nutrition, Hospital Universitario Ramón y Cajal, Universidad de Alcalá, Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS)
Locations (1):
- Lía Nattero Chávez, Madrid, Please Select, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nattero-Chavez L, de La Calle E, Lecumberri-Pascual E, Bayona Cebada A, Ruiz Gracia T, Quintero Tobar A, Lorenzo Monino M, Sanchez Rodriguez C, Izquierdo A, Escobar-Morreale HF, Luque-Ramirez M. Comparing quality of life in traditional face-to-face visits with a hybrid approach of telemedicine with in-person follow-ups in recent users of advanced closed-loop systems: a randomized controlled clinical trial in patients with type 1 diabetes. Ther Adv Endocrinol Metab. 2024 Oct 25;15:20420188241288789. doi: 10.1177/20420188241288789. eCollection 2024. PMID 39493410
- [Derived] Nattero-Chavez L, Lecumberri Pascual E, De La Calle E, Bayona Cebada A, Ruiz T, Quintero Tobar A, Lorenzo M, Sanchez C, Izquierdo A, Luque-Ramirez M, Escobar-Morreale HF. Switching to an advanced hybrid closed-loop system in real-world practice improves hypoglycemia awareness and metabolic control in adults with type 1 diabetes, particularly in those with impaired perception of hypoglycemia symptoms. Diabetes Res Clin Pract. 2023 May;199:110627. doi: 10.1016/j.diabres.2023.110627. Epub 2023 Mar 20. PMID 36940793